CLINICAL TRIAL: NCT06150014
Title: Randomized, Double-blind, Placebo-controlled Phase Ib/IIa Clinical Trial to Evaluate the Efficacy and Safety of TQA3605 Tablets Monotherapy or in Combination With Nucleoside (Acid) Analogues in Treatment-naïve Patients and Treated Patients With Chronic Hepatitis B
Brief Title: A Clinical Study of TQA3605 Tablets Monotherapy or in Combination With Nucleoside (Acid) Analogues in Treatment Naive and Treated Patients With Chronic Hepatitis B
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA3605-Ib/IIa-01
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Placebo +Nucleoside (acid) analogs (NAs) combination therapy 24 weeks (Placebo Comparator): Placebo and Nucleoside (acid) analogues, taken orally once daily, continue for 24 weeks.
  Interventions: Drug: Placebo; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 50 mg of TQA3605 tablets +NAs combination therapy 24 weeks (Active Comparator): 50 mg of TQA3605 tablets and Nucleoside (acid) analogues, taken orally once daily, continue for 24 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 100 mg of TQA3605 tablets +NAs combination therapy 48 weeks (Active Comparator): TQA3605 is taken orally 100mg once daily; Nucleoside (acid) analogues were used once daily for 48 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 200 mg of TQA3605 tablets +NAs combination therapy 48 weeks (Active Comparator): TQA3605 is taken orally 200mg once daily; Nucleoside (acid) analogues were used once daily for 48 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- Placebo +Nucleoside (acid) analogs (NAs) combination therapy (Placebo Comparator): Placebo taken orally once daily, continue for 12 weeks. Placebo was then combined with nucleoside (acid) analogues (once daily) for 36 weeks
  Interventions: Drug: Placebo; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 100 mg of TQA3605 tablets +NAs combination therapy (Active Comparator): TQA3605 was taken orally 100mg once a day for 12 weeks. It was then combined with nucleoside (acid) analogues (once daily) for 36 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 200 mg of TQA3605 tablets +NAs combination therapy (Active Comparator): TQA3605 was taken orally 200mg once a day for 12 weeks. It was then combined with nucleoside (acid) analogues (once daily) for 36 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet
- 300 mg of TQA3605 tablets+NAs combination therapy (Active Comparator): TQA3605 was taken orally 300mg once a day for 12 weeks. It was then combined with nucleoside (acid) analogues (once daily) for 36 weeks.
  Interventions: Drug: TQA3605 tablets; Drug: Entecavir dispersible tablets; Drug: Tenofovir disoproxil fumarate tablet; Drug: Tenofovir alafenamide fumarate tablet

INTERVENTIONS:
Drug: Placebo — TQA3605 placebo tablets were orally administered on an empty stomach (at least 2 hours before or after meals) with warm.
  Arms: Placebo +Nucleoside (acid) analogs (NAs) combination therapy; Placebo +Nucleoside (acid) analogs (NAs) combination therapy 24 weeks
Drug: TQA3605 tablets — TQA3605 inhibits viral replication.
  Arms: 100 mg of TQA3605 tablets +NAs combination therapy; 100 mg of TQA3605 tablets +NAs combination therapy 48 weeks; 200 mg of TQA3605 tablets +NAs combination therapy; 200 mg of TQA3605 tablets +NAs combination therapy 48 weeks; 300 mg of TQA3605 tablets+NAs combination therapy; 50 mg of TQA3605 tablets +NAs combination therapy 24 weeks
Drug: Entecavir dispersible tablets — Entecavir inhibits viral replication and indicated for chronic hepatitis B treatment.
Drug: Tenofovir disoproxil fumarate tablet — Tenofovir disoproxil fumarate is a Nucleotide reverse transcriptase inhibitor.
Drug: Tenofovir alafenamide fumarate tablet — Tenofovir alafenamide fumarate inhibits hepatitis B virus replication.

SUMMARY:
A randomized, double-blind Phase Ib/IIa multicenter trial design was used. All eligible subjects received TQA3605 tablets/placebo plus nucleoside (acid) analogues. A total of 88 subjects were required

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Male and female, ≥18 years old and ≤70 years old (subject to the date of signing the informed consent);
* Patients diagnosed with chronic hepatitis B (CHB) who have been serum HBsAg positive for more than 6 months and HBeAg positive or negative ;
* The liver fibrosis ultrasound transient imaging elastic technology (Fibroscan/FibroTouch) showed that the liver hardness (LSM) was less than 12.4 Kpa;
* Patients with chronic hepatitis B after treatment;
* Treatment-naïve patients of chronic hepatitis B patients;

Exclusion Criteria:

* Complicated with other infected disease such as hepatitis A virus (HAV), hepatitis C virus (HCV), Hepatitis D virus (HDV), hepatitis E virus (HEV), human immunodeficiency virus (HIV), syphilis (syphilis antibody positive and need treatment determined by the investigator);
* Abdominal ultrasound or other imaging or histology showed suspected cirrhosis or other liver disease before or during screening;
* Patients have a history of hepatocellular carcinoma (HCC) before or at the time of screening, or may be at risk for HCC;
* Active autoimmune disease diagnosed with immunodeficiency or undergoing systemic therapy which was continuing within 2 weeks before first dosing;
* Currently being treated with nephrotoxic drugs or drugs that alter renal excretion;
* Abnormal thyroid function;
* Renal diseases such as chronic kidney disease and renal insufficiency or creatinine clearance (CLCr) <60 ml/min during the screening period;
* Hematologic and biochemical abnormalities;
* History of allergy to the investigational drug or its excipients;
* Recipients of solid organs or bone marrow transplants;
* A history of malignant tumors within the past 5 years;
* Interstitial lung disease, acute lung disease, etc.;
* Uncontrolled systemic diseases such as high blood pressure and diabetes;
* Have used any investigational drug or participated in a clinical trial within one month prior to the administration of study drug;
* Those who received live attenuated vaccine within 28 days before the start of study treatment, inactivated vaccine within 7 days, or planned vaccination during the study period;
* The investigator determines that there is any medical or psychiatric condition that puts the subject at risk, interferes with participation in the study, or interferes with the interpretation of the study results;
* Female subjects that were pregnant, lactating or had a positive pregnancy result during the screening period or during the trial; Male and female patients with reproductive potential who were unwilling to use effective contraceptive methods during the study period;
* Subjects who have any medical condition that may affect the absorption of oral drugs;
* Within 12 weeks prior to screening, treated chronic hepatitis B patients who had stopped taking nucleoside (acid) analogues for more than 14 consecutive days;
* Those considered unsuitable for enrollment by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) | Up to 48 weeks
  The incidence of adverse events (AEs) during treatment
Severity of adverse events (AEs) | Up to 48 weeks
  The severity of adverse events (AEs) during treatment
Incidence of serious adverse events (SAEs) | Up to 48 weeks
  The incidence of serious adverse events (SAEs) during treatment
Severity of serious adverse events (SAEs) | Up to 48 weeks
  The severity of serious adverse events (SAEs) during treatment

SECONDARY OUTCOMES:
Incidence of abnormal laboratory test values | Up to 48 weeks
  The incidence of abnormal laboratory values during treatment, e.g. triglycerides.
Severity of abnormal laboratory test values | Up to 48 weeks
  The severity of abnormal laboratory values during treatment, e.g. triglycerides.
Deoxyribonucleic acid level of hepatitis B virus | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  Changes in hepatitis B virus deoxyribonucleic acid (HBV DNA) levels from baseline
Hepatitis B surface antigen | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  Changes in serum hepatitis B surface antigen (HBsAg) from baseline
Hepatitis B e antigen | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  Changes in serum hepatitis B e antigen (HBeAg) from baseline
Serologic clearance and/or serologic conversion of HBsAg | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  Proportion of subjects with HBsAg serologic clearance and/or serologic conversion
Serologic clearance and/or serologic conversion of HBeAg | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  Proportion of subjects with HBeAg serologic clearance and/or serologic conversion
Virological breakthrough rate | At week 12, week 24, week 36 and week 48 or when subjects withdrawal from the study
  The proportion of subjects who achieved a virological breakthrough (defined as a confirmed increase of HBV DNA levels >1.0 log10 IU/ml from the minimum during treatment).
Peak time (Tmax) | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  Time to reach peak blood concentration after a single dose
Peak concentration | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The highest plasma drug concentration that can be achieved after medication
Area under blood concentration-time curve (AUC) | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The amount of drug absorbed into the human circulation after a single dose can be estimated using the area under the blood concentration-time curve
Apparent volume of distribution (Vd/F) | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  When a drug reaches homeostasis in the body, the ratio of the amount of drug in the body to the blood concentration is called the apparent volume of distribution.
Plasma clearance | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The amount of plasma that the kidneys completely clear in unit time (per minute).
Elimination half-life | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The time it takes for the plasma concentration to drop by half.
Steady state peak time | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The time required to reach peak steady-state concentration after administration
Steady state maximum concentration | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The highest blood concentration that occurs after stabilization
Steady state minimal concentration | pre-dose, 30 minutes, 1 , 2 , 4 , 6 , 12, 24 hours after administration on Day 1; pre-dose on Day 8 and Day 9; pre-dose, 30 minutes, 1, 2, 4, 6, 12, 24 hours after administration on Day 10.
  The lowest blood concentration that occurs after stabilization

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of the Chinese People's Liberation Army Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi